CLINICAL TRIAL: NCT01379157
Title: The Pharmacodynamics of Imipenem in Critically Ill Patients With Ventilator-associated Pneumonia Following Administration by 4 h or 0.5 h Infusion
Brief Title: Pharmacodynamics Study of Imipenem in Patients With Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Prof.Dr.Sutep Jaruratanasirikul, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISP 39337
Record Dates: First submitted 2011-05-05; First posted 2011-06-23 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2011-12

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Patients with ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Imipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional arm (Active Comparator): Infusion of 0.5 g of imipenem for 0.5 hr every 6 hr for 3-5 days
  Interventions: Drug: Imipenem
- Extended infusion arm (Experimental): Infusion of 1 g of imipenem for 4 hr every 8 hr for 3-5 days
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Imipenem — Each patient will receive a loading dose of 0.5 g 3 min infusion followed by 0.5 hr infusion of 0.5 g every 6 hr of imipenem at room temperature
  Other Names: Tienam
  Arms: Conventional arm
Drug: Imipenem — Each patient will receive a loading dose of 0.5 g 3 min infusion followed by 4 hr infusion of 1 g every 8 hr of imipenem at room temperature
  Other Names: Tienam
  Arms: Extended infusion arm

SUMMARY:
Imipenem is a carbapenem antibacterial agent with a broad spectrum of activity against Gram-negative and Gram-positive bacteria. This agent is often used as the last line of therapy for highly resistant Gram negative bacilli nosocomial infections. In common with other beta-lactamase inhibitor, the main pharmacokinetic/pharmacodynamic (PK/PD) index that correlates with the therapeutic efficacy is the time that concentrations in the tissue and serum are above the MIC and administration by continuous infusion is the preferred mode of administration to maximize this parameter.

However, in tropical countries, the stability of carbapenem antibiotics is an important consideration when considering continuous infusion. Therefore, prolonged infusion may be a useful mode of administration to maximize bactericidal activity. This study will demonstrate the stability of imipenem in clinical use at room temperature in tropical countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > or = 20 years
* Patients who have VAP with Gram negative bacilli infections which are sensitive to imipenem by the disk diffusion

Exclusion Criteria:

* Patients who have documented hypersensitivity to imipenem or other carbapenems
* Patients who have an estimated creatinine clearance of < or = 60 ml/min
* Patients who are in circulatory shock
* Patients who are pregnant

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Accessed PK/PD parameters | 24 hours profile after first dose of trail drug.
  - To determine plasma Imipenem PK/PD parameters (the PK/PD index (T>MIC), the probability of target attainment (PTA) at 40% (T>MIC), the cumulative fraction of response (CFR))after 4 hr infusion of 1 gm every 8 hr compared to 0.5 hr infusion of 0.5 gm every 6 hr.
  Conventional arm: after first dose, blood samples will be obtained by direct venepuncture at: time 0, 0.5, 6, 6.5, 12, 12.5, 18, 18.25, 18.5, 18.75, 20, 21, 22 and 24 hr Extended infusion arm: after first dose, blood samples will be obtained by direct venepuncture at: time 0, 4, 8, 12, 16, 16.5, 17, 18, 20, 20.5, 21, 22, and 24 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand